CLINICAL TRIAL: NCT03720015
Title: Concurrent Training and Nutritional Management Prevent Body Weight Loss During Radiotherapy in a Young Adult With Head and Neck Cancer: A Case Control Study
Brief Title: Concurrent Training and Nutritional Management in Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, Luis Berlanga, Principal Investigator, Universidad Francisco de Vitoria
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0003
Record Dates: First submitted 2018-10-16; First posted 2018-10-25 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Body Weight Changes
MeSH Terms: conditions — Body Weight Changes | interventions — Exercise; Diet

STUDY DESIGN:
Intervention Model Description: Case study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent training (Experimental): Three sessions per week of concurrent training during radiotherapy period. Each session will begin with warm-up (5-min cardiovascular activity at low-moderate intensity, joint mobility and one set of resistance exercises circuit at 30-40% 1RM). Resistance training will follow the warm-up, including 9 standard exercises involving major muscle groups of the lower and upper body: vertical bench press, parallel bar dip for triceps, seated rowing, standing dumbbell curl for biceps, leg press, deadlift and shoulder press. All these exercises will be realized following circuit training with 4 sets of 8-12 repetitions, using a training load of 70-80% RM. When patient will able to complete more than 12 repetitions, load will be increased progressively 10%. Cardiovascular training will be completed 20-30 min after resistance training, and it will include High-Intensity Interval Training (HIIT) of 3 min near to the second ventilatory threshold and 2 min near to the first ventilatory threshold.
  Interventions: Behavioral: Physical exercise
- Nutritional management (Experimental): Prescribed diet controlling macronutrients according to patient body weight (~4g/kg/day for carbohidrates, ~2g/kg/day for proteins, and ~1g/kg/day for fats). Patient will take one single dosage per day of probiotics (Arkoprobiotics® Defenses), 1 or 2 capsules of omega-3 fish oil concentrate (Solgar®, 600-1200mg depending on fat sources intake during the day), and a combine ingestion of 3g beta-hydroxybeta-methylbutyrate (HMB), 14g arginine, and 14g glutamine (HSN Raw Series®, all pure ingredients and making the ingestion adding each of them individually in a solution with 300-400 ml of water). During concurrent training sessions, between resistance exercise and HIIT, patient will also take 6g of BCAA's (HSN Raw Series®, 2:1:1) along with a banana. Additionally, patient could take whey isolated protein (Amix® IsoPrime CFM) to meet with some of the prescribed proteins intakes.
  Interventions: Dietary Supplement: Nutritional management

INTERVENTIONS:
Behavioral: Physical exercise — Physical exercise controlled program supervised by an accredited exercise specialist
  Arms: Concurrent training
Dietary Supplement: Nutritional management — Nutritional management controlled by a PhD clinical and sport nutrition specialist
  Arms: Nutritional management

SUMMARY:
A case control study with before-after design. A concurrent training and a nutritional management intervention was offered by a patient with head and neck cancer, in order to compare outcomes related to strength and endurance performance and to body composition

DETAILED DESCRIPTION:
Cancer causes important public health problems around the world and it is one of the most frequent cause of death overall. Among non-pharmacological treatment, physical exercise has shown improvements in different types of cancer and patients, but it is important to define the optimal dose. Our aim is to determine the effects of a concurrent training program and a nutritional management developed during radiotherapy treatment on physical performance and body composition. A patient with an oral cavity cancer will develop three sessions per week of concurrent training: resistance training included 9 standard exercises involving major muscle groups (4x8-12 RM), and cardiovascular training included a High-Intensity Interval Training (HIIT). Nutritional management will include a diet controlling macronutrients (~4g/kg/day for carbohidrates, ~2g/kg/day for proteins, and ~1g/kg/day for fats), along with some nutritional supplements such as beta-hydroxybeta-methylbutyrate (HMB), arginine, glutamine, omega-3 fish oil concentrate, and BCAA's during training sessions. Intervention took place during radiotherapy period (7 weeks). We expect that body composition will remain invariable, and 1RM will increased. VO2max is expected to be almost the same, but intensity tolerated at maximum VO2max could be higher. If our results confirm that, we could conclude that a combination between resistance exercise and HIIT along with a nutritional management developed during radiotherapy could be effective to prevent muscle mass loss and muscle function decrease in a young patient with oral cavity cancer.

ELIGIBILITY:
This is a case control study

Ages: 32 Years to 34 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-09-17 (Actual)

PRIMARY OUTCOMES:
Body weight in kilograms (kg) | 8 weeks
Total fat in percentage (%) | 8 weeks
Lean body mass in percentage (%) | 8 weeks
Visceral adipose tissue in cm2 | 8 weeks

SECONDARY OUTCOMES:
1 repetition maximal (1RM) for upper-body in kilograms (kg) | 8 weeks
  Test will be performed in vertical bench press
1 repetition maximal (1RM) for lower-body in kilograms (kg) | 8 weeks
  Test will be performed in leg press
Maximal oxygen uptake (VO2max) in ml/kg/min | 8 weeks
  Test will be performed in a cycloergometer
Power at VO2max in watts (W) | 8 weeks
  Test will be performed in a cycloergometer

CONTACTS AND LOCATIONS:
Locations (1):
- Francisco de Vitoria University (UFV), Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided